CLINICAL TRIAL: NCT05034302
Title: Posture Analysis Through Machine Learning
Acronym: PathML
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: SentiMetrix, Inc (Industry)
Collaborators: California Polytechnic State University-San Luis Obispo (Other)
Responsible Party: Principal Investigator, Vadim Kagan, President, SentiMetrix, Inc
Other Study IDs: PathML2021
Record Dates: First submitted 2021-08-27; First posted 2021-09-05 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Health Behavior
Keywords: adult; behavioral observation; methodology; computer vision
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Recordings: Selection criteria include individuals between the ages of 18-85 years, no major chronic illness that impair mobility and able to complete activities of daily living without assistance. We will recruit approximately equal number of men and women and 30% of the sample will be racial or ethnic minorities.

SUMMARY:
This study will include video-recorded data from 20 adults (age 18-85yrs) residing in San Luis Obispo, CA. Participants will also have their height and weight measured, complete demographic questionnaires, and one 3hour session with video recordings in a combination of naturalistic condition and semi-structured environments. The video data will be used to train machine learning models to automatically classify physical behavior as compared to ground-truth measures of manual annotation.

DETAILED DESCRIPTION:
This is a cross-sectional, single observation study. Individuals will be drawn from local surrounding clinics and the general community. All recruitment will include both men and women. Selection criteria include individuals between the ages of 18-85 years, no major chronic illness that impair mobility and able to complete activities of daily living without assistance. Participants will complete one three hour session where there will be one video camera set up within the home (i.e., static cameras). For approximately 30 minutes of the session they will complete a semi-scripted routine that will include sit to stand transitions, a timed up and go test, and scripted activities of daily living.

Researchers will use a video camera to record participant behavior within their daily life. For two of the three hours, researchers will be video recordings the participants normal (unscripted) activities. • For one hour of the session we will use two cameras, one that will be held by a researcher and one that will be set up on a tripod. During this hour we will ask participants to follow a semi-structured protocol:

* 10 minutes recording the empty space
* 10 minutes that include a timed up a go test (sit up from a chair and walk 10 feet), repeat the test 3 times.
* 6 minute walk test (walk continuously for 6 minutes)
* Four stage balance test
* The remainder of the time, participants will complete standard activities of daily living like household chores, eating or drinking.

Data will be annotated using an established behavioral observation software by training research assistants (ground-truth). The image data from videos will be used to train machine learning models to classify physical activities (e.g. ,'walking', 'sitting' or 'standing up"), information about behavior (e.g., location and purpose of the activity), and performance (e.g., walking speed and sit to stand transition times).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-85 years
2. No major chronic illness that impair mobility
3. Able to complete activities of daily living without assistance.

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Generally health adult population recruited from local community
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Postural Status | Upon enrollment (one timepoint)
  Sitting versus standing versus moving
Activity type | Upon enrollment (one timepoint)
  Indoor vs outdoor vs driving
Sit to stand transition time | Upon enrollment (one timepoint)
  Time it takes to go from sitting to standing

SECONDARY OUTCOMES:
Activity intensity | Upon enrollment (one timepoint)
  Sedentary, light, moderate and vigorous intensity
Activity type | Upon enrollment (one timepoint)
  lying, sitting, driving, standing, housework or office work, walking, running, sports, other

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Keadle, Principal Investigator — Cal Poly
Locations (1):
- CalPoly, San Luis Obispo, California, United States

IPD SHARING:
Plan to Share IPD: No